CLINICAL TRIAL: NCT00637741
Title: Physician Initiated Trial Investigating the Efficacy of the Implant of EverFlex 200mm Long Nitinol Stents in TASC C&D Femoropopliteal Lesions
Brief Title: DURABILITY-200: EverFlex 200mm Long Nitinol Stents in TASC C&D Femoropopliteal Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Flanders Medical Research Program (FMRP), Flanders Medical Research Program (FMRP)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-004
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Peripheral Vascular Disease; Intermittent Claudication; Critical Limb Ischemia
Keywords: Peripheral Vascular Disease; Intermittent claudication; Critical Limb Ischemia; TASC
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everflex 200 (Experimental): study group treated with at least one 200 mm Everflex stent
  Interventions: Device: Everflex 200

INTERVENTIONS:
Device: Everflex 200

SUMMARY:
The objective of this clinical investigation is to evaluate the long-term (up to 12 months) outcome of the 200 mm long self-expanding nitinol EverFlex (ev3) stent in long femoropopliteal lesions (TASC C & D) Is is the first time that the use of 200 mm long stents will be evaluated in these lesions. It is expected that the outcome of the treatment with this type of long stents will be better as the treatment of identical lesions lengths with multiple shorter stents.

ELIGIBILITY:
Inclusion Criteria:

GENERAL

* De novo, restenotic or reoccluded lesion located in the femoropopliteal arteries suitable for stenting
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Prior to enrollment, the guidewire has crossed target lesion
* Patient is eligible for treatment with the self-expanding nitinol EverFlex (ev3) stent

ANGIOGRAPHIC

* The target lesion is located within the native femoropopliteal artery until maximally 3 cm proximally of the knee joint.
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* The target lesion, visually estimated, has a minimal length of 15 cm and can be categorized as either a type C or D lesions according the TASC II guidelines
* Target vessel diameter visually estimated is >4mm and <6.5 mm
* There is angiographic evidence of at least one-vessel-runoff to the foot

Exclusion Criteria:

* Presence of another stent in the target vessel that was placed during a previous procedure
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Previous by-pass surgery in the same limb
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Aneurysm located at the level of the SFA
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Ipsilateral iliac treatment before the target lesion procedure with a residual stenosis > 30% or ipsilateral iliac treatment conducted after the target lesion procedure
* Use of thrombectomy, artherectomy or laser devices during procedure
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary patency defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without TLR | 12 months

SECONDARY OUTCOMES:
Technical success, defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex imaging. | procedure
Primary patency defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without TLR | 6 months
Clinical success at follow-up defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure | 6 & 12 months
Stent fracture rate determined on x-ray (Mild - single strut fracture; Moderate - fracture of more than one strut but without complete separation; Severe - complete separation) | 12 months
Serious adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint-Blasius, Dendermonde, Belgium
Locations (2):
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde

REFERENCES:
- [Derived] Bosiers M, Deloose K, Callaert J, Moreels N, Keirse K, Verbist J, Peeters P. Results of the Protege EverFlex 200-mm-long nitinol stent (ev3) in TASC C and D femoropopliteal lesions. J Vasc Surg. 2011 Oct;54(4):1042-50. doi: 10.1016/j.jvs.2011.03.272. Epub 2011 Jun 2. PMID 21636239